CLINICAL TRIAL: NCT06938971
Title: Effects of Exercise Training on Health-related Quality of Life in Patients With Unresectable Metastatic Colorectal Cancer: A Multi-center Randomized Controlled Trial
Brief Title: Randomized Controlled Trial of the Effects of Combined Resistance and AerobiC Exercise on Health-related Quality of Life in Patients Undergoing First-line Chemotherapy for Metastatic Colorectal Cancer (REACH)
Acronym: REACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Casper Simonsen, Group Leader, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Exercise mCRC
Record Dates: First submitted 2025-03-31; First posted 2025-04-22 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
Keywords: Exercise; Physical activity; Metastatic colorectal cancer; Colorectal cancer; Endurance training; Oncology; Chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity; Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants allocated to the control group will receive standard care. No restrictions regarding physical activity will be imposed.
- Exercise training (Experimental): Participants allocated to the exercise intervention group will receive standard care plus an exercise intervention. The exercise intervention will of consist moderate-to-high intensity supervised and unsupervised home-based exercise training (bicyling, walking, or running) 5 times/week for 18 weeks.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Participants allocated to the exercise intervention group will receive standard care plus an exercise intervention. The exercise intervention will consist moderate-to-high intensity supervised and unsupervised home-based exercise training (bicyling, walking, or running) 5 times/week for 18 weeks.
  Arms: Exercise training

SUMMARY:
The primary objective of this trial is to compare the effects of 18 weeks structured exercise training versus on control on healt-related quality of life in patients with unresectable mCRC.

ELIGIBILITY:
Inclusion criteria:

- Adults (≥18 years of age) schduled to undergo chemotherapy for the treatment of unresectable metastatic colorectal cancer.

Exclusion criteria :

* Pregnancy.
* A life expectancy of < 6 months.
* Absolute contraindications to maximal exercise, as per the recommendations by the Danish Society of Cardiology.
* ECOG (Eastern Cooperative Oncology Group) performance status > 2.
* Inability to understand the Danish or English language.
* Engagement in structured moderate-to-high aerobic exercise training for >30 min >1 times/week for the past 3 months at the time of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | Every 3 weeks from randomization until post-intervention (18 weeks), withdrawal of consent to participate, or death (whichever occurs first)
  The difference in means of the average global health-related quality of life score in intervention versus control, regardless of intervention compliance; disease progression; cancer treatment discontinuation or dose-modifications; changes in initially scheduled cancer treatment; and engagement in alternative cancer care, in physical activity, structured exercise training, or municipality-based cancer rehabilitation. Health-related quality of life will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30. Scores range from 0 to 100, with higher scores indicating better health-related quality of life.

SECONDARY OUTCOMES:
Health-related quality of life | Randomization and 3, 6, 9, 12, 15, and 18 weeks after randomization or until withdrawal of consent to participate, or death (whichever occurs first). Followed-up at 36, 52, 104, and 156 weeks after randomization.
  The difference in means of the average health-related quality of life score (global score and score for each subcomponent) in intervention versus control, regardless of intervention compliance; disease progression; cancer treatment discontinuation or dose-modifications; changes in initially scheduled cancer treatment; and engagement in alternative cancer care, in physical activity, structured exercise training, or municipality-based cancer rehabilitation. Health-related quality of life will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30. Scores range from 0 to 100.
Colorectal cancer-specific symptoms | Randomization and 3, 6, 9, 12, 15, and 18 weeks after randomization or until withdrawal of consent to participate, or death (whichever occurs first). Followed-up at 36, 52, 104, and 156 weeks after randomization.
  The difference in means of the average colorectal cancer-specific symptoms inter-vention versus control, regardless of intervention compliance; disease pro-gression; cancer treatment discontinuation or dose-modifications; changes in initially scheduled cancer treatment; and engagement in alternative can-cer care, in physical activity, structured exercise training, or municipality-based cancer rehabilitation. Health-related quality of life will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire CR 29. Scores range from 0 to 100.
Cancer related fatigue | Randomization and 3, 6, 9, 12, 15, and 18 weeks after randomization or until withdrawal of consent to participate, or death (whichever occurs first). Followed-up at 36, 52, 104, and 156 weeks after randomization.
  Between-group difference in changes in cancer related fatigue from randomization to 6, 12, 18, 36, 52, 104, and 156 weeks after randomization. Cancer related fatigue will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core FA12. Scores range from 0 to 100.
Patient-reported symptomatic adverse events | 7 days after every second cycle of treatment, starting from the second cycle. Each cycle is 2-3 weeks, depending on the regimen.
  Patient-reported symptomatic adverse events will be assessed, using the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). A total of 42 symptomatic adverse events have been preselected based on high expected prevalence in patients with colorectal cancer.
Serious adverse events | From randomization to 20 weeks after randomization
  Serious adverse events.
Unscheduled hospitalizations | From randomization to 20 weeks after randomization
  Unscheduled hospitalizations.
Dose delays of chemotherapy | From randomization to 20 weeks after randomization
  A chemotherapy dose delay is a delay of the planned administation of chemotherapy.
Dose reductions of chemotherapy | From randomization to 20 weeks after randomization
  A chemotherapy dose reduction is a decrease of the planned dose of chemotherapy.
Discontinuation of chemotherapy | From randomization to 20 weeks after randomization
  Discontinuation of chemotherapy is a premature discontinuation of the planned chemotherapy.
Estimated maximal oxygen uptake | Randomization, 18 weeks after randomization
  Between-group difference in changes from randomization to 18 weeks after randomization. Maximal oxygen uptake (mL/kg/min) will be estimated from ratings of perceived exertion obtained during submaximal exercise.
Estimated maximal oxygen uptake | Randomization, 18 weeks after randomization
  Between-group difference in changes from randomization to 18 weeks after randomization. Maximal oxygen uptake (L/min) will be estimated from ratings of perceived exertion obtained during submaximal exercise.
Hand-grip strength | Randomization, 18 weeks after randomization
  Between-group difference in changes from randomization to 18 weeks after randomization. Handgrip strength (kg) of the dominant hand will be measured using a dynamometer
Balance | Randomization, 18 weeks after randomization
  Between-group difference in changes from randomizationto 18 weeks after randomization. Standing balance will be assessed using side-by-side stands, semi-tandem stands, and tandem stands. The time until the participants move their feet or grasp for support will be measured. The test is terminated after 10 seconds. Balance will be scored in accordance with the standardized scoring guidelines of the Short Physical Performance Battery (SPPB).
Habitual 4 m Gait Speed | Randomization, 18 weeks after randomization
  Between-group difference in changes from randomization to 18 weeks after randomization. Habitual 4 m gait speed will be measured on a 4 m straight, flat walking course and scored in accordance with the standardized scoring guidelines of the Short Physical Performance Battery (SPPB).
Chair Rising Capacity | Randomization, 18 weeks after randomization
  Between-group difference in changes from randomizationto 18 weeks after randomization. Chair rising capacity will be assessed using a sit-to-stand test. The time taken to perform five stands will be measured and scored in accordance with the standardized scoring guidelines of the Short Physical Performance Battery (SPPB).
Short Physical Performance Battery (SPPB) total score | Randomization, 18 weeks after randomization
  Between-group difference in changes from randomization to 18 weeks after randomization. The Short Physical Performance Battery (SPPB) total score will be calculatedin accordance with the standardized scoring guidelines of the SPPB.
Lean mass | Randomization, 18 weeks after randomization
  Between-group difference in changes from randomization to 18 weeks after randomization. Whole-body lean mass (kg) will be measured using bioelectrical impedance analysis.
Fat mass | Randomization, 18 weeks after randomization
  Between-group difference in changes from randomization to 18 weeks after randomization. Whole-body fat mass (kg) will be measured using bioelectrical impedance analysis.
Body mass | Randomization, 18 weeks after randomization
  Between-group difference in changes from randomizationto 18 weeks after randomization. Body mass (kg) will be measured using an electronic scale.
Body mass index | Randomization, 18 weeks after randomization
  Between-group difference in changes from randomizationto 18 weeks after randomization.
Resting heart rate | Randomization, 18 weeks after randomization
  Between-group difference in changes from randomization to 18 weeks after randomization. Reported as beats/min.
Systolic blood pressure | Randomization, 18 weeks after randomization
  Between-group difference in changes from randomizationto 18 weeks after randomization. Reported as mmHg.
Diatolic blood pressure | Randomization, 18 weeks after randomization
  Between-group difference in changes from randomizationto 18 weeks after randomization. Reported as mmHg.
3-year overall survival | From randomization to 3 years after randomization
  Overall survival, defined as the time from randomization to death.
3-year progression-free survival, defined as the time from randomization to disease progression or death | From randomization to 3 years after randomization
  3-year progression-free survival, defined as the time from randomization to disease progression or death.
Time to progression, defined as the time from randomization to disease progression | From randomization to 3 years after randomization
  Time to progression, defined as the time from randomization to disease progression
Time to treatment failure | From randomization to 3 years after randomization
  Time to treatment failure, defined as the time from initiation of treatment to early discontinuation.
Proportion of participants undergoing intended curative surgery from randomization to post-intervention. | From randomization to 20 weeks after randomization
  Proportion of participants undergoing intended curative surgery.

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Centre for Physical Activity Research, Copenhagen Univerisity Hospital - Rigshospitalet, Copenhagen
  - Herlev and Gentofte Hospital, Herlev
  - North Zealand University Hospital, Hillerød, Hillerød
  - Zealand University Hospital, Roskilde, Roskilde

IPD SHARING:
Plan to Share IPD: Undecided